CLINICAL TRIAL: NCT07011043
Title: A Phase 1b Open-Label, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Budoprutug (TNT119) in Adult Subjects With Systemic Lupus Erythematosus (SLE)
Brief Title: A Phase 1b Study of Budoprutug in Systemic Lupus Erythematosus (SLE)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Climb Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TNT119-SLE-101
Record Dates: First submitted 2025-05-06; First posted 2025-06-08 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus; SLE; Biologics; Open-label; Monoclonal; Anti-CD19
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Intervention Model Description: This is an open-label study in which subjects will be enrolled into four single-dose ascending cohorts. Each subject's participation will last approximately 198 days, including a 30-day screening period, a 1-day treatment period, and follow-up through Week 24.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Dose Level A (Experimental)
  Interventions: Drug: Budoprutug
- Cohort 2: Dose Level B (Experimental)
  Interventions: Drug: Budoprutug
- Cohort 3: Dose Level C (Experimental)
  Interventions: Drug: Budoprutug
- Cohort 4: Dose Level D (Experimental)
  Interventions: Drug: Budoprutug

INTERVENTIONS:
Drug: Budoprutug — Single IV dose of study product on Day 1 of study
  Other Names: TNT119

SUMMARY:
The main objective is to assess the safety and tolerability of budoprutug in adults with SLE. Pharmacokinetics, pharmacodynamics, and preliminary clinical efficacy will also be assessed.

DETAILED DESCRIPTION:
Budoprutug is a humanized, immunoglobulin (Ig) G1 monoclonal antibody that selectively binds to CD19 and is projected to deplete targeted cells through antibody-dependent cellular cytotoxicity. This Phase 1b, open-label study will evaluate budoprutug administered as a single intravenous infusion in ascending dose cohorts of patients aged 18 years and above with active, seropositive SLE and inadequate response to standard therapy. The study will also assess the pharmacokinetics, pharmacodynamics and early indications of efficacy of budoprutug in SLE, where pharmacodynamics will be evaluated as the change in the number of B cells and immunoglobulins (antibodies) in the blood over time following a single infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 65 years at the time of consent.
2. Diagnosis of SLE according to the 2019 European League Against. Rheumatism and the American College of Rheumatology (ACR) classification criteria.
3. Active, seropositive disease, with SLEDAI 2K >=8.
4. Inadequate response to at least 2 therapeutic interventions, including at least one oral immunosuppressive or biologic standard-of care therapy.

Exclusion Criteria:

1. Active neuropsychiatric SLE.
2. History of inflammatory or autoimmune diseases including, but not limited to, rheumatoid arthritis, scleroderma, myositis, vasculitis, inflammatory bowel disease, or other conditions that require immune suppressive therapy. Subjects with stable concurrent Sjogren's, asthma, or autoimmune thyroid disease may be considered for participation.
3. Active systemic infection or history of chronic, recurrent, latent, or recent serious infections.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) | Up to Week 24
  Number of participants experiencing TEAEs, graded per NCI CTCAE v5.0.
Incidence of Clinical Laboratory Abnormalities | Up to Week 24
  Number of participants with clinically significant laboratory abnormalities.
Change from Baseline in Systolic Blood Pressure | Up to Week 24
  Mean change from baseline in systolic blood pressure (mmHg).
Change from Baseline in Diastolic Blood Pressure | Up to Week 24
  Mean change from baseline in diastolic blood pressure (mmHg).
Change from Baseline in Heart Rate | Up to Week 24
  Mean change from baseline in heart rate (bpm).
Change from Baseline in Respiratory Rate | Up to Week 24
  Mean change from baseline in respiratory rate.
Change from Baseline in Body Temperature | Up to Week 24
  Mean change from baseline in body temperature (°C).
Change from Baseline in PR Interval | Up to Week 24
  Mean change from baseline in PR interval (ms).
Change from Baseline in QRS Duration | Up to Week 24
  Mean change from baseline in QRS duration (ms).
Change from Baseline in QT Interval | Up to Week 24
  Mean change from baseline in QT interval (ms).
Change from Baseline in QTc Interval | Up to Week 24
  Mean change from baseline in corrected QT interval (QTc).

SECONDARY OUTCOMES:
Area Under the Curve (AUC) of Budoprutug | Up to Week 24
  Measurement of the area under the drug concentration-time curve.
Maximum Observed Plasma Concentration (Cmax) | Up to Week 24
  Measurement of the maximum observed plasma concentration.
Time to Maximum Observed Concentration (Tmax) | Up to Week 24
  Measurement of the time to maximum observed concentration.
Terminal Half-Life (T1/2) | Up to Week 24
  Measurement of the terminal half-life in days.
Apparent Clearance (CL/F) of budoprutug | Up to Week 24
  Measurement of the apparent clearance in L/hour.
Volume of Distribution (Vd) | Up to Week 24
  Measurement of the volume of distribution in liters.
Change from Baseline in Circulating B Cell Count | Up to Week 24
  Change in absolute number of CD19+ B cells in peripheral blood.
Incidence of Anti-Drug Antibodies (ADAs) | Up to Week 24
  Number of participants with detectable ADAs.
ADA Titer Over Time | Up to Week 24
  Measurement of ADA titer over time.

OTHER OUTCOMES:
Change from Baseline in BILAG-2004 Score | Up to Week 24
  Measurement of change in BILAG-2004 score from baseline.
Change from Baseline in SLEDAI-2K Score | Up to Week 24
  Measurement of change in SLEDAI-2K score from baseline.
Change from Baseline in Physician's Global Assessment | Up to Week 24
  Measurement of change in Physician's Global Assessment score from baseline.
Proportion of Participants Achieving SRI-4 Response | Up to Week 24
  Percentage of participants achieving SRI-4 response.
Change from Baseline in Urine Protein Creatinine Ratio (UPCR) | Up to Week 24
  Measurement of change in UPCR from baseline.
Time to Renal Response | Up to Week 24
  Measurement of time to renal response in weeks.
Proportion of Participants with Complete or Partial Renal Response | Up to Week 24
  Percentage of participants with complete or partial renal response.
Change from Baseline in FACIT-Fatigue Score | Up to Week 24
  Measurement of change in FACIT-Fatigue score from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Climb Bio, Inc.
Locations (18):
- United States (2):
  - Climb Bio Investigative Site #100104, Allen, Texas
  - Climb Bio Investigative Site #100101, San Antonio, Texas
- Bulgaria (2):
  - Climb Bio Investigative Site# 359101, Plovdiv
  - Climb Bio Investigative Site# 359102, Sofia
- Georgia (2):
  - Climb Bio Investigative Site #995102, Tbilisi
  - Climb Bio Investigative Site #995101, Tbilisi
- Greece (2):
  - Climb Bio Investigative Site# 300102, Exochi, Thessaloniki
  - Climb Bio Investigative Site# 300103, Thessaloniki, Thessaloniki
- Climb Bio Investigative Site #100103, Caguas, Puerto Rico
- Climb Bio Investigative Site# 400101, Cluj-Napoca, Romania
- Spain (2):
  - Climb Bio Investigative Site# 340101, Sabadell, Barcelona
  - Climb Bio Investigative Site# 340102, A Coruña
- Ukraine (6):
  - Climb Bio Investigative Site #380102, Ivano-Frankivsk
  - Climb Bio Investigative Site #380103, Kyiv
  - Climb Bio Investigative Site #380106, Kyiv
  - Climb Bio Investigative Site #380101, Ternopil
  - Climb Bio Investigative Site #380104, Vinnytsia
  - Climb Bio Investigative Site #380105, Vinnytsia